CLINICAL TRIAL: NCT05635123
Title: A Cohort Study of Uterine Malignancies
Status: Recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20220352-R
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and surgical tissue samples （cancers） were collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — This is a prospective observational study with no intervention.

SUMMARY:
The purposes of current study were to explore the relationship between cervical cancer/endometrial cancer and demographic information, behavior and life style, pregnancy-related factors, and disease history, and to study the factors affecting the prognosis of cancers. In addition, omics tests were performed on the biological specimens to identify the diagnostic markers and prognostic biomarkers.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients who meet the eligibility requirements will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years;
* Women with cervical cancer or endometrial cancer with a definite pathological diagnosis for the first time;
* Women attending a health check-up;
* Obtain informed consent and sign an informed consent form.

Exclusion Criteria:

* Patients who are unable to cooperate with the investigations such as mental disorders or cognitive impairment；
* Patients with cancer other than cervical cancer or endometrial cancer;
* Women who have received hysterectomy or pelvic radiation therapy previously.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators establish a population cohort of 6200 women including patients with cervical cancer or endometrial cancer, and women attending to a health check-up.
Sampling Method: Non-Probability Sample
Enrollment: 6200 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 60 months
  progression free survival for patients with cervical cancer or endometrial cancer

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, PhD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's hospital school of medicine zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No